CLINICAL TRIAL: NCT02186366
Title: Study of Abdominal Massage Therapy for Generalized Anxiety Disorder Based on the " Essence Fosters Spirit " Theory
Brief Title: Efficacy Study of Abdominal Massage Therapy to Treat Generalized Anxiety Disorder of Deficiency of Both Heart and Spleen Type
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Qing (Other)
Responsible Party: Sponsor-Investigator, Sun Qing, deputy director of the Tuina Department, First Teaching Hospital of Tianjin University of Traditional Chinese Medicine
Organization: First Teaching Hospital of Tianjin University of Traditional Chinese Medicine (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TECF 20120210
Record Dates: First submitted 2014-06-23; First posted 2014-07-10 (Estimated); Last update posted 2014-09-03 (Estimated); Status verified 2014-09

CONDITIONS: Anxiety Disorders
Keywords: Anxiety Disorders, Massage Therapy, Treatment Efficacy
MeSH Terms: conditions — Anxiety Disorders | interventions — Buspirone

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Abdominal Massage Therapy (Experimental): Abdominal Massage Therapy , 30 minutes, three times one week for 6 weeks
  Interventions: Drug: Buspirone
- Buspirone (Active Comparator): Buspirone by mouth 5mg three times per day for 6week
  Interventions: Other: Abdominal Massage Therapy

INTERVENTIONS:
Other: Abdominal Massage Therapy — Abdominal Massage Therapy , 30 minutes, three times one week for 6 weeks. If the subjects have recovered in the treatment of 6 weeks, we can end treatment early.
  Other Names: Abdominal Tuina Manipulation
  Arms: Buspirone
Drug: Buspirone — Buspirone by mouth 5mg three times per day for 6week. If the subjects have recovered in the treatment of 6 weeks, we can end treatment early.
  Other Names: Buspirone HCl
  Arms: Abdominal Massage Therapy

SUMMARY:
Generalized Anxiety Disorder (GAD) is characterized by the presence of persistent worry or fear of no explicit object and fixed content, or things that might occur in real life，which not corresponds with the realities. Patients with GAD may occur a series of somatic symptoms including muscle tension, backaches, headaches, fatigue, insomnia, restlessness, as well as psychological feelings of anxiety, worry and feeling overwhelmed. And it always brings some type of functional disability or decrease in quality of life. GAD is treated by Selective Serotonin Reuptake Inhibitors (SSRIs) or Serotonin, Norepinephrine Reuptake Inhibitors(SNRI) and 5-ht1a receptor agonists as regular medication which have the definite effects. But, some adverse reaction of SSRIs or SNRI leads to the compliance of taking medicine of patients with GAD. There is an impressive data suggesting that Abdominal Massage Therapy is effective in decreasing some symptoms of somatic symptoms and psychological feelings.

This study is designed as a parallel group, positive control, non-inferiority study. It will recruit 140 cases of generalized anxiety disorder of deficiency of both heart and spleen type. Both the treatment group and the control group will be randomly assigned 70 cases. Patients in the treatment group will be treated by Abdominal Massage for 6 weeks，and the control group by buspirone . The total study includes 4 views that are respectively before the treatment，after 3 weeks treatment, after the whole treatment , and 3 months after the whole treatment. At all of the 4 views, all participants will be estimated the scores of Hamilton Depression Scale(HAMD) ,self-rating anxiety scale(SAS), and Quality of life assessment scale. At the second, third and the forth views, all participants will be estimated Clinical Global Impression ( CGI). At the first and the third views, all participants will be collected the data of content of hydroxytryptamine（5-HT）, Norepinephrine and total cortisol in blood plasma, and of blood stream speed, vascular resistance index and pulsatility index of middle cerebral artery （MCA）, anterior cerebral artery（ACA）, posterior cerebral artery （PCA） and basilar artery（BA）. This study aims to investigate the efficacy of Abdominal Massage Therapy vs. buspirone, and discover the correlation between these scales and these objective indicators.

DETAILED DESCRIPTION:
Quality control: The study site and all researchers must comply with the required qualifications. All researchers must be trained before the study. The study will take a number of measures to ensure the recruitment of the required sample size, and compliance of intervention providers and participants.

ELIGIBILITY:
Inclusion Criteria:

* Meet criteria for a primary diagnosis of current GAD as demonstrated by a structured clinical interview for Diagnostic and Statistical Manual -IV（DSM-IV）；meet a diagnosis of Deficiency of both heart and spleen type.
* The scores of SAS≥50, 24≥the scores of HAMD ≥15.
* The symptoms of anxiety have continued not less than 6months.

Exclusion Criteria:

* major depression, schizophrenia ,bipolar disease other psychotic disorders, drug-dependent persons;
* patients with severe suicidal tendencies;
* women in pregnancy or breastfeeding, menstrual or postpartum recovery;
* suffered from serious illness or impairment of system,such as heart and brain blood vessels, lungs, liver, kidneys and blood system.
* persons allergic to Buspirone and excipient;
* persons suffering from epilepsy or hypertension or Glaucoma or myasthenia gravis or leukopenia;
* persons must be taking monoamine oxidase inhibitors;
* persons who drink a lot;
* persons with the local skin lesions in abdomen damage (such as damage, Burns, etc);
* persons with abdominal visceral tumors, nodules, inflammation, edema, abdominal aortic atherosclerosis;
* persons without the incompetence or unable to read, write and understand independently;
* persons whom the researchers believe should not participate in this study.

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 140 (Estimated)
Dates: Start 2014-09; Primary Completion 2015-10 (Estimated)

PRIMARY OUTCOMES:
reductive rate of Hamilton Depression Scale（ HAMD reductive rate） | baseline and post- 6week intervention
  We will estimate the scores of the Hamilton Depression Scale of participants at baseline and post- 6week intervention，then calculate the HAMD reductive rate according to the following formula：HAMD reductive rate=（scores of HAMD at baseline - scores of HAMD at post- 6week intervention ）/ scores of HAMD at baseline×100%

SECONDARY OUTCOMES:
Scores of Hamilton Depression Scale(HAMD) | baseline, post- 3week intervention, post- 6week intervention and post-3month after 6- week intervention
  We will estimate the scores of the Hamilton Depression Scale of participants.
Scores of self-rating anxiety scale( SAS) | baseline, post- 3week intervention, post- 6week intervention and post-3month after 6- week intervention
  We will estimate the scores of the self-rating anxiety scale of participants.
Scores of Quality of life assessment scale | baseline, post- 3week intervention, post- 6week intervention and post-3month after 6- week intervention
  We will estimate the scores of the Quality of life assessment scale of participants.
Scores of Clinical Global Impression | post- 3week intervention and post- 6week intervention and post-3month after 6- week intervention
  We will estimate the scores of Clinical Global Impression.

OTHER OUTCOMES:
content of 5-HT in blood plasma | baseline and post- 6week intervention
  We will test the content of 5-HT of participants in blood plasma and record the data.
content of Norepinephrine in blood plasma | baseline and post- 6week intervention
  We will test the content of Norepinephrine of participants in blood plasma and record the data.
content of total cortisol in blood plasma | baseline and post- 6week intervention
  We will test the content of total cortisol of participants in blood plasma and record the data.
blood stream speed of MCA, ACA, PCA and BA | baseline and post- 6week intervention
  We will test blood stream speed of MCA, ACA, PCA and BA of patients by Transcranial Doppler and record the data.
vascular resistance index of MCA, ACA, PCA and BA | baseline and post- 6week intervention
  We will test vascular resistance index of MCA, ACA, PCA and BA of patients by Transcranial Doppler and record the data.
pulsatility index of MCA, ACA, PCA and BA | baseline and post- 6week intervention
  We will test pulsatility index of MCA, ACA, PCA and BA of patients by Transcranial Doppler and record the data.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Tianjin University of Traditional Chinese Medicine, Tianjin, Tianjin Municipality, China